CLINICAL TRIAL: NCT04802473
Title: "Influence of Flap Thickness Upon Root Coverage With the Use of Acellular Dermal Matrix: a Prospective Case Series"
Brief Title: Flap Thickness Upon Root Coverage With the Use of Acellular Dermal Matrix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Jose Nart Molina, Chairman and Program Director, Department of Periodontology UIC-Barcelona, Universitat Internacional de Catalunya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PER-ECL-2019-06
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Gingival Recession; Periodontal Attachment Loss; Periodontal Diseases; Soft Tissue Injuries
MeSH Terms: conditions — Gingival Recession; Periodontal Attachment Loss; Periodontal Diseases; Soft Tissue Injuries

STUDY DESIGN:
Intervention Model Description: A prospective case series with a 6-month follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gingival recession treatment (Experimental): Gingival recession treatment by means of tunnel technique and OrACell dermal matrix.
  Interventions: Procedure: Mucogingival surgery

INTERVENTIONS:
Procedure: Mucogingival surgery — In brief description, Tunnel+acellular dermal matrix treatment will be performed by starting initial sulcular incisions, tunneling knives will be used to elevate the buccal gingiva by means of a full-thickness flap elevation. Flap preparation will be extended beyond the MGJ. The exposed root surfaces will be treated with pre-conditioning EDTA (Straumann PrefGel®) for 2 minutes. ADM (OrACELL, LifeNet Helth, Virginia Beach, VA, USA) of 1.25-1.75mm in thickness will be cut to the exact size of the defect, and will be inserted into the tunnel, and subsequently covered advancing the flap by means of sling sutures to stabilize the flap in a coronal position (6-0 Polypropylene, Prolene, Ethicon, Johnson and Johnson, New Brunswick, NJ, USA). Sutures will be removed after 14 days. Two weeks after surgery, patients will resume mechanical tooth cleaning with a soft toothbrush. Patients will be recalled at 1, 3 and 6 months for professional oral hygiene procedures.
  Other Names: Treatment of adjacent multiple gingival recessions using the OrACell® dermal matrix

SUMMARY:
OrACell has been tested as a barrier in bone regenerative procedures showing promising results in new bone formation after socket preservation, but no data is available on root coverage procedures. Moreover, it has been suggested that keratinized tissue width (KTW) ≥2mm and gingival thickness (GT) ≥1.2 mm at 6 months of the surgical procedures are two important predictors for long term stability of gingival margin Therefore, it was hypothesized that soft tissue thickness and keratinized tissue width may influence the percentage of root coverage. By means of a prospective case series (12 patients in total), the aim is to study the performance of the OrACell dermal matrix in the treatment of multiple and adjacent gingival recessions, determining the amount of complete root coverage obtained at 6 months of follow-up. At the same time, it is intended to evaluate the effect of initial gingival thickness, by means of digital scanning, upon the success of root coverage procedure with OrACell.

DETAILED DESCRIPTION:
Background:

Gingival recession is a lesion characterized by clinical attachment loss of the periodontal apparatus to the root surface of the tooth, resulting in an apical migration of the gingival margin that occasionally generates esthetic problems, hypersensitivity and difficulty in maintaining proper hygiene. To correct this, the additional use of connective tissue grafts in root coverage procedures has reported highly predictable results. Over time, different substitutes such as acellular dermal matrix (ADM), xenografts (XEN) have been suggested to reduce patient morbidity by avoiding the donor site. Recently, an acellular dermal allograft known as OrAcell® has shown good results in terms of soft tissue regeneration and guided bone/tissue regeneration.

Objectives:

Overall objective The objective of this prospective case series is to evaluate the influence of initial soft tissue thickness (STT) upon the success of a surgical root coverage procedure Specific objective To assess the statistical correlation of keratinized tissue width (KTW) and VD on the outcome (%RC) of the TUN plus acellular dermal matrix (ADM).

Hypothesis:

Null hypothesis H01: STT is not a predictor for root coverage procedures and does not influence the percentage of root coverage.

H02: KTW is not a predictor for root coverage procedures and does not influence the percentage of root coverage.

H03: VD is not a predictor for root coverage procedures and does not influence the percentage of root coverage.

Alternative hypothesis:

H11: STT is a predictor for root coverage procedures and detrimentally influences the percentage of root coverage.

H12: KTW is a predictor for root coverage procedures and a low VD detrimentally influences the percentage of root coverage.

H13: VD is a predictor for root coverage procedures and detrimentally influences the percentage of root coverage.

Material and methods:

Study design This is a prospective case series with a 6-month follow-up.

Setting of the study The study will be performed at a private practice setting associated to the Universitat Internacional de Catalunya (UIC). Subjects will be selected, on a consecutive basis, among individuals referred to a specialist periodontist's private practice.

Study population:

Subjects affected by at least one GR in single rooted teeth will be included in the study. They will be selected, on a consecutive basis, among individuals referred to the authors private practice. The study protocol and informed consent will be reviewed by the Ethical Committee of the Universitat Internacional de Catalunya, Barcelona, Spain and will be conducted the Helsinki Declaration, 1975, as revised in 2013.

Surgical treatment:

All surgeries will be performed by expert periodontists (GB). In brief description, TUN+ADM treatment will be performed by starting initial sulcular incisions, tunneling knives will be used to elevate the buccal gingiva by means of a full-thickness flap elevation. Flap preparation will be extended beyond the MGJ. The periosteum will be cut, and a blunt dissection into the vestibular lining mucosa will be carried out to eliminate muscle tension so that the mucosal flap can be passively positioned above the level of CEJ on the teeth. The exposed root surfaces will be treated with pre-conditioning EDTA (Straumann PrefGel®) for 2 minutes. ADM (OrACELL, LifeNet Helth, Virginia Beach, VA, USA) of 1.25-1.75mm in thickness will be cut to the exact size of the defect, and will be inserted into the tunnel, and subsequently covered advancing the flap by means of sling sutures to stabilize the flap in a coronal position (6-0 Polypropylene, Prolene, Ethicon, Johnson and Johnson, New Brunswick, NJ, USA).

Patients will be instructed to avoid any mechanical trauma or toothbrushing in the surgical sites for 2 weeks. Analgesic medication (ibuprofen) will be prescribed as required and patients will be instructed to rinse with Chlorhexidine three times per day for 2 weeks. Sutures will be removed after 14 days. Two weeks after surgery, patients will resume mechanical tooth cleaning with a soft toothbrush. Patients will be recalled at 1, 3 and 6 months for professional oral hygiene procedures.

Post-surgical instructions and infection control:

Patients will be instructed to avoid any mechanical trauma or tooth brushing in the surgical sites for 2 weeks. Analgesic medication (ibuprofen) will be prescribed as required and patients will be instructed to rinse with Chlorhexidine 0.12% two times per day for 2 weeks. Sutures will be removed after 14 days. Two weeks after surgery, patients will resume mechanical tooth cleaning with a soft toothbrush. Patients will be recalled at 1, 3 and 6 months for professional oral hygiene procedures.

Blindness The clinical examiner (RP) will be unaware of digital measurements performed by a second researcher (JV) and vice versa.

Blindness will be maintained strictly confidential by the investigators.

Data collection:

A guidebook will be prepared to systematize the procedures for sample and data collection. The data will be later transferred to a computerized database (Epidata®, Odense, Denmark, Europe).

A) Sociodemographic data An interview will be conducted during the pre-surgical visit to obtain information regarding age, sex, medical history, use of medication, exposure to tobacco, pregnancy and previous periodontal surgeries.

B) Clinical measurements The following clinical measurements will be performed by blinded examiners () using a periodontal probe (PCP UNC 15, Hu-Friedy, Chicago, IL, USA): Probing Depth PD and keratinized tissue width (KTW). KTW will be measured at the most apical point in the GM to the mucogingival junction at the mid-buccal site to the nearest millimeter. KTT will be measured 1.5mm and 3mm apical to the GM using an injection needle, perpendicular to the tissues surface and a silicon stop over the gingival surface and fixed with a cyanoacrylic adhesive ().

C) Digital measurements A digital scan of the arch with the teeth to be treated will be performed with an optical 3D measurement system (3Shape Trios®, Copenhagen, Denmark) creating Surface Tessellation Language (STL) files. The acquired data will be transferred into a digital imaging software (3Shape Trios®, Erlangen, Germany). Baseline and corresponding follow-up scans of each clinical case will be then virtually superimposed and matched into one common coordinate system (Geomagic, 3D Systems, Research Triangle Park, NC, USA) using the tool Control X. By using the buccal surfaces of the concerned teeth as reference points for the superpositioning of the different time points (pre-operative and post-operative), this approach will allow for precise evaluation of dimensional soft tissue alterations over time by a blinded examiner (JV).

The following measurements will be taken:

* RD will be measured from CEJ to the GM in a cross section at the central buccal site (24).
* Change in KTT will be measured as mean thickness of the marginal soft tissues by superimposing STL files at 1.5mm and 3mm apical to the GM.

All clinical measurements and volumetric evaluations of the soft will be performed at baseline, 3 months and at 6 months after surgery.

D) Patient reported outcomes measures (PROMS)

Patient reported outcomes in terms of aesthetics and morbidity during treatment will be evaluated as follows:

A total of seven questions will be evaluated at suture removal using a visual analogue scale (VAS score; VAS 0-100, 100 reflecting the highest morbidity). Pain during surgery, pain and swelling in the weeks following the mucogingival surgery until suture removal will be assessed for the recipient site. Patients will be further asked about their willingness to repeat the treatment. In addition, the use of pain medication and the number of days pain medication taken will be reported at the same time- point.

Moreover, patients' esthetic satisfaction will be recorded by means of a visual analog scale (VAS) with a score between 0 (poor) and 10 (excellent).

Withdrawal of consent The Patient Information Sheet will clearly state that the patient can withdraw from the study at any time without prejudice or explanation. Such withdrawal will be documented in the medical record file.

Sample size calculation The study is powered based on an objective of this study, the correlation between the outcome of root coverage (%MRC) and an anatomical independent continuous variable, the STT. A previous study (25) reported a statistically significant negative correlation between root prominence and linear root coverage measurements (r= -0.8). Using this data and accepting an alpha risk of 5%, a beta risk of 10% in a one-sided test and assuming a 10% of dropout, a minimum of 12 patients/sites were determined as necessary to conduct the research.

Due to the methodological discrepancies regarding the surgical approach and the primary with the aforementioned article (25) an interim analysis will be performed to reassess statistical power and determine the need of increasing or not the sample size.

Statistical analysis:

Descriptive statistics will be calculated for continuous and categorical variables using means and standard deviations or frequencies and percentages, respectively.

Data distribution will be assessed by means of Shapiro Wilk test. Differences between baseline, 3 and 6 months post-operatively quantitative variables will be analyzed using a generalized lineal model or Friedman test according to the distribution of the variables. With regard to qualitative variables, McNemar test will be performed to compare differences between groups.

The association or correlation between CRC and % of CRC and STT will be evaluated using he Pearson or Spearman correlation coefficient.

MRC will be calculated using the following formula: [(preoperative RD) - (postoperative RD))/(preoperative RD)] x 100. The RC% will be transformed to a binary variable (the presence of 100% of complete RC [CRC]). At each timepoint logistic multilevel models, considering both patient and tooth levels, will be performed to investigate factors influencing the CRC. Baseline variables will be included in the models as explicative variables.

The level of statistical significance will be set at p <.05. Analysis will be performed by the use of SPSS 22.0 software package (IBM SPSS, SPSS Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Periodontally and systemically healthy.
* Presence of Cairo RT 1 and RT2 GR defects
* Recession ≥2mm in depth at the buccal aspect.
* Full-mouth plaque and bleeding score ≤20%.
* No previous periodontal surgery.
* Presence of identifiable CEJ (a step ≤1mm at the CEJ and/or presence of root abrasion, but with identifiable CEJ, will be accepted).

Exclusion Criteria:

* Tobacco smoking of ≥10 cigarettes a day.
* Contraindications for periodontal surgery.
* Medications known to affect the gingiva or interfere with wound healing.
* Pregnancy.
* Active orthodontic therapy.
* Caries or restorations in the area to be treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Complete root coverage (CRC) | CRC 6 months after surgery
  By using the buccal surfaces of the concerned teeth as reference points for the superpositioning of the different time points (pre-operative and post-operative), this approach will allow for precise evaluation of dimensional soft tissue alterations over time by a blinded examiner

SECONDARY OUTCOMES:
: Mean Root Coverage (MRC), change in Keratinized tissue width and change in Keratinizedd tissue thickness | 6 months after surgery
  By using the buccal surfaces of the concerned teeth as reference points for the superpositioning of the different time points (pre-operative and post-operative), this approach will allow for precise evaluation of dimensional soft tissue alterations over time by a blinded examiner

CONTACTS AND LOCATIONS:
Overall Officials: Jose Nart, PhD, Principal Investigator — UIC
Locations (1):
- Gonzalo Blasi, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No